CLINICAL TRIAL: NCT06816732
Title: The Effect of Nurse-led Modular Training on Self-efficacy and Disease Adaptation in Patients Diagnosed With Hypertension
Brief Title: The Effect of Modular Education on Individuals Diagnosed With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulviye Özcan Yüce (Other)
Responsible Party: Sponsor-Investigator, Ulviye Özcan Yüce, Assistant Professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-59754796-050.99-65645
Record Dates: First submitted 2025-01-20; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: Hypertension; nursing; self-efficacy; modular training; adaptation to chronic illness
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: A pre-test post-test, randomized-controlled research method
Masking Description: Blinding was impossible because the research involved a training program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modular training (Experimental): The intervention group participants filled out all the data collection tools in the first interview and three months later. They received modular training by phone 2 weeks, 4 weeks, 8 weeks, and 12 weeks after the first interview.
  Interventions: Behavioral: Nurse-led Modular Training
- Control (No Intervention): The control group participants filled out all the data collection tools in the first interview and three months later. They did not receive any modular training.

INTERVENTIONS:
Behavioral: Nurse-led Modular Training — The intervention group participants filled out all the data collection tools in the first interview and three months later. They received modular training by phone 2 weeks, 4 weeks, 8 weeks, and 12 weeks after the first interview.The modular training addressed (1) defining hypertension, (2) systemic effects of hypertension, (3) general effects of antihypertension drugs, (4) regular medication and blood pressure monitoring, and (5) eating a healthy diet and being active (what to do for a better heart health and a more stable blood pressure)
  Arms: Modular training

SUMMARY:
Aim:This study focused on patients with hypertension to investigate the effect of a nurse-led counseling program on their self-efficacy and disease adherence.

DETAILED DESCRIPTION:
This study adopted a randomized-controlled and intervention research method. Data were collected between September 2022 and February 2023 at the internal medicine outpatient clinic of Adana City Hospital.

Participants were recruited using random sampling. Simple randomization was used to allocate both groups equally and randomly (https://www.randomizer.org/). The researcher first created a randomization list. Then, she assigned participants to the intervention and control groups according to the list. Blinding was impossible because the research involved a training program. A power analysis (G*Power 3.1.9.4) was performed based on the effect size (d = 0.93) reported by Zhang et al. (Zhang et al., 2021). The results showed that a sample of 62 would be large enough to detect significant between-group differences (power 95%, margin of error 5%, and confidence interval 95%). The results showed that a sample of 42 was large enough to detect significant differences [alpha= 0.05 and power (1- beta) 0.80]. However, each group comprised 23 participants to avoid missing data and the execute parametric tests.Data were collected using a personal information form, the Hypertension Self-Efficacy Scale (HSES), the Modified Morisky Scale (MMS), and the Adaptation to Chronic Illness Scale (ACIS). The inclusion criteria were (1) having had hypertension at least for six months, (2) being an adult (over 18), (3) not having received training on hypertension before, (4) having no communication problems, (5) not being pregnant, and (6) volunteering.

ELIGIBILITY:
Inclusion Criteria:

* Having had hypertension at least for six months
* Being an adult (over 18),
* Not having received training on hypertension before,
* Having no communication problems,
* Not being pregnant,
* Volunteering

Exclusion Criteria:

* Hypertension diagnosis duration is less than 6 months
* Having verbal communication problems
* Not volunteering to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Effect of nurse-led modular training program on self-efficacy of individuals diagnosed with hypertension | 3 months
  It is expected that the pre-training self-efficacy scale score averages of the patients in the intervention group will increase after the training. For this purpose, the Hypertension Self-efficacy Scale was used. Self-Efficacy Scale in Hypertension was used to determine the self-efficacy levels of patients diagnosed with hypertension. The scale consists of 20 items. The items of the scale are in the 4-point Likert type, ranging from "not at all appropriate" (1 point) to "very appropriate" (4 points). The total score of the scale varies between 20-80 points. An increase in the total score obtained from the scale indicates an increase in the level of self-efficacy in hypertension.
Effect of nurse-led modular education program on hypertensive individuals' adaptation to disease | 3 months
  It is aimed that the average score of the patients in the intervention group on the chronic disease adaptation scale before the training will increase after the training.For this purpose, the chronic disease adjustment scale was used.The Scale of Adjustment in Chronic Diseases is a 5-point Likert type and consists of 25 items and three sub-dimensions: physical adjustment, social adjustment and psychological adjustment. The scale ranges from 1 (strongly disagree) to 5 (strongly agree). Negative items are reverse scored. The highest score is 125. An increase in the score obtained from the scale indicates a high level of patient adjustment to the disease.
Effect of nurse-led modular education program on medication motivation of individuals diagnosed with hypertension | 3 months
  The Turkish Modified Morisky Scale was used to test this. The Turkish Modified Morisky Scale is a reliable, easy-to-apply scale consisting of six questions that can separately evaluate the knowledge and motivation levels regarding drug use habits. In the evaluation of the answers given as "Yes" or "No"; the yes answer to the 2nd and 5th questions was calculated as 1 point, the no answer as 0 points; and the yes answer to the other questions was calculated as 0 points, the no answer as 1 point. The total score received by the patient from the 1st, 2nd and 6th questions; 0 or 1 indicates a low motivation level, while values above 1 indicate a high motivation level. The total score received from the 3rd, 4th and 5th questions; 0 or 1 indicates a low knowledge level, and values above 1 indicate a high knowledge level.
Effect of a nurse-led modular education program on medication motivation of individuals diagnosed with hypertension | 3 months
  Turkish Modified Morisky Scale (Moriskiy motivation level) was used to evaluate the effect of the nurse-led modular training program on medication motivation of individuals diagnosed with hypertension.This scale questions the belief in the benefit of the treatment, the habit of taking the medications on time, and the situation of forgetting or stopping to take the medication. In the evaluation of the answers given as "Yes" or "No"; the yes answer to the 2nd and 5th questions was calculated as 1 point, the no answer as 0 points; and the yes answer to the other questions was calculated as 0 points, the no answer as 1 point. The total score received by the patient from the 1st, 2nd and 6th questions; 0 or 1 indicates a low motivation level, while values above 1 indicate a high motivation level. The total score received from the 3rd, 4th and 5th questions; 0 or 1 indicates a low knowledge level, and values above 1 indicate a high knowledge level.

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Turkey (Türkiye)